CLINICAL TRIAL: NCT02774408
Title: Effects of Automated Adjustment of Inspired Oxygen With Combined Adaptive Mechanical Backup Ventilation as Compared to Automated Oxygen Adjustment Alone in Preterm Infants With Intermittent Hypoxemic Events During Non-invasive Ventilatory Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ulm (Other)
Collaborators: Dr. von Hauner Children's Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Helmut Hummler, Professor, University of Ulm
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FiO2 Backup
Record Dates: First submitted 2016-03-24; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Apnea, Hypoxia
Keywords: backup ventilation; preterm infants; functional residual capacity; chronic lung disease
MeSH Terms: conditions — Apnea; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Other): Infants on CPAP will receive backup breafs whenever the SpO2 <88 % along with
  automated FiO2 controller. In the control period they will receive automated FiO2
  alone
  Interventions: Device: Saturation sensitive backup ventilation
- NIMV/NIPPV (Other): Infants on NIMV NIPPV will receive an increase in the backup rate to 2 times the rate
  of the backup triggered by apnoe (apnoe time 5s), whenever the SpO2 under 88%
  ( max rate 100/min) in the reference period as compared to baseline (automated FiO2
  - control + unchanged SIPPV settings)
  Interventions: Device: Saturation sensitive backup ventilation

INTERVENTIONS:
Device: Saturation sensitive backup ventilation

SUMMARY:
In this 2-phase cross-over study the investigators test the hypothesis that automated adjustment of the inspired oxygen with the combined use of synchronized noninvasive SpO2-sensitive and apnea-sensitive backup-ventilation (S-NIPPV) increases the time within the intended oxygen saturation range as compared to automated FiO2 adjustment alone.

DETAILED DESCRIPTION:
This study will be a randomized-controlled clinical study with cross-over design of two treatment phases of 24h duration each (1. Automated FiO2-adjustment (SPO2C), 2. combined use of automated FiO2-adjustment and SpO2-sensitive/apnea-sensitive S-NIPPV (SPO2C + BU), see Figures 1 and 2). The investigators will study two patient groups of premature infants depending on the type of respiratory support at study time: One group, where the infants are on CPAP at study time, and another group of preterm infants who are already supported by nasopharyngeal IPPV at study time. Both studies will be sufficiently powered to show a significant treatment effect if it is present. Study infants will be recruited in the neonatal ICU of the children's hospital, University of Ulm and the neonatal ICU, University of Munich. Both NICU team have participated previously in clinical trials investigated new modes of mechanical ventilation using automated ventilation adjustment in the target population.

Randomization of the sequence of the two study phases will be carried out using sealed envelopes. Infants will be changed to a specific ventilator device approved for clinical use in neonates in Germany (Sophie®-Respirator, Stephan Medizintechnik GmbH, Gackenbach, Germany), which is capable to automatically adjust the FiO2 (called "SPO2C") and to apply noninvasive backup-ventilation (using a noninvasive trigger device (S-NIPPV) or non-synchronized nasal IPPV (NIPPV) based on readings of an incorporated SpO2 monitoring device (Masimo® Radical 7, averaging time 2 sec). Synchronization of NIPPV and detection of apnea is achieved by using the Graseby capsule (Stephan, Vio Healthcare Ltd, Ref. 103560103), which will be secured onto the anterior abdominal wall near to the right costal margin.

Infants on CPAP (first group) will be exposed to the first study phase (SPO2C, or SPO2C + BU, Figure 1) for 24h and then will be switched to the alternate mode for 24h each. Infants, who are already on nasal IPPV (SIPPV or NIPPV) as chosen by the clinical team will be exposed to NIPPV with a standardized inflation rate of 40 breaths/min (nonsynchronized, because this seems to be the current standard of care according to the available literature) and SPO2C, or to SPO2C plus synchronized BU (starting with a rate of 80 inflations/min with stepwise weaning) and then will be switched to the alternate mode for 24h each.

ELIGIBILITY:
Inclusion Criteria:

1. postmenstrual age <34 wks GA at study time (<32 wks GA at birth)
2. on nasal/nasopharyngeal CPAP or nasal IMV / IPPV
3. at least 4 desaturations (SpO2 <80%) during an 8 hour period within the 24h before the study using a standard pulse oximeter incorporated in the NICU (Masimo SET, Irvine, CA, averaging time 8 sec; delay 10s)
4. informed consent obtained from the parents or legal guardian

Exclusion Criteria:

1. postnatal age <96h (to exclude rapidly changing conditions during the early phase of RDS and to avoid handling of the infant during the critical period for IVH)
2. congenital cyanotic heart disease
3. no decision for full treatment support
4. Average FiO2 during the last 24h bevor the active study phase >0.60 (too sick for non-invasive ventilator support)
5. Congenital malformations of the lung or the diaphragm (i.e. diaphragmatic hernia, congenital cystic lung diseases...)
6. Clinical evidence for seizures
7. Ongoing Sepsis with hemodynamic compromise (defined as a CrP > 20mg/l or positive blood culture (for sepsis), and requirement of catecholamines (for hemodynamic compromise))
8. Need of blood-transfusion during study time

Ages: 96 Hours to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the total duration of time with an arterial oxygen saturation as measured by pulse oxymetry (percentage of the total recording time) within the target range (88-95%). | 48 hours

SECONDARY OUTCOMES:
the number of episodes with an SpO2 <80% | 48 hours
The number of extended/very long episodes outside the SpO2 target range (defined as episodes with a duration of more than 1 minute/3 minutes) | 48 hours
Mean SpO2. | 48 hours
Variability of SpO2 (coefficient of variation) | 48 hours
Mean FiO2 during the study time | 48 hours
The workload for the medical staff as measured by the number of manual adjustments of FiO2 because of episodes of hyperoxemia | 48 hours
The workload for the medical staff as measured by the number of manual adjustments of FiO2 because of episodes of hypoxemia. | 48 hours
Tissue oxygenation measurement (measured with near infrared spectrometry) of different organs (kidney, brain, muscle ) | 48 hours

OTHER OUTCOMES:
the number of episodes with an SpO2 <80%. | 48hours
the number of episodes with an SpO2 <70%. | 45hours
the mean duration of episodes with an SpO2 with hyperoxemia (SpO2 >96%). | 48hours
The mean duration of episodes with an SpO2 <80% | 48 hours